CLINICAL TRIAL: NCT03545867
Title: Effect of Various Forms of Upper Body Exercise on the Energetic Response to a Meal in Persons With Spinal Cord Injury
Brief Title: Energetic Response to Feeding and Exercise in SCI
Acronym: CRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20171114
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injuries
Keywords: postprandial; glycemia; lipemia; macronutrient metabolism; physical activity
MeSH Terms: conditions — Spinal Cord Injuries; Hyperlipidemias; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Static first arm with randomized remaining three arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Seated control (CON) (Experimental): Participants remain seated in their habitual wheel chair for ~45 min (duration of exercise performed in other arms). Following the intervention they are fed.
  Interventions: Behavioral: Seated control (CON); Other: Liquid Meal
- Circuit resistance training (CRT) (Experimental): Participants complete upper extremity resistance maneuvers (lifts) interspersed with low-load/high-speed arm cycling for a combined 30 repetitions of 6 lifts and ~20 min of arm cycling. During this time energy expenditure is measured via open-circuit indirect calorimetry. Following the intervention they are fed.
  Interventions: Behavioral: Circuit resistance training (CRT); Other: Liquid Meal
- Moderate intensity continuous (MICT) (Experimental): Participants complete continous arm cycling at a steady-state power output (intensity) matched to the energy expenditure (kcal/min) and duration of exercise (min) response during CRT. Following the intervention they are fed.
  Interventions: Behavioral: Moderate intensity continuous (MICT); Other: Liquid Meal
- High intensity interval training (HIIT) (Experimental): Participants complete interval arm cycling at power output that varies between 2 min "active" and two min "recovery" periods. This interval exercise is matched to the total energy expenditure (accumulated kcals) response during CRT. Following the intervention they are fed.
  Interventions: Behavioral: High intensity interval training (HIIT); Other: Liquid Meal

INTERVENTIONS:
Behavioral: Seated control (CON) — Seated rest
  Arms: Seated control (CON)
Behavioral: Moderate intensity continuous (MICT) — Arm cycling at a continuous power output
  Arms: Moderate intensity continuous (MICT)
Behavioral: High intensity interval training (HIIT) — Arm cycling at power outputs that vary between high and low intensity intervals
  Arms: High intensity interval training (HIIT)
Behavioral: Circuit resistance training (CRT) — Alternating between six upper extremity resistance maneuvers interspersed with low-resistance/high-speed arm cycling.
  Arms: Circuit resistance training (CRT)
Other: Liquid Meal — A liquid meal consisting of 600 kcal comprised of 50% carbohydrate, 35% fat, and 15% protein (by kcal).

SUMMARY:
This study investigates the effect of various forms of upper extremity exercise on postprandial glycemia and lipemia in persons with spinal cord injury (SCI). Participants are measured at rest and fed a standardized meal following seated rest (CON), moderate intensity continuous arm cycling (MICT), high intensity interval arm cycling (HIIT), and circuit resistance exercise (CRT) matched for exercise energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>/=18 years of age)
* Neurologically stable chronic (>/= 1year) spinal cord injury (SCI)
* American Spinal Injury Association Impairment Scale (AIS) grade A, B, or C
* SCI at level </= the first thoracic vertebrae (T1)

Exclusion Criteria:

* Being of ≤ 18 years of age.
* Contraindication to exercise (ACSM Guideline, 10th edition)
* Lower extremity fracture or dislocation within 6 months of participation,
* History head injury or seizures.
* Inability to consent.
* Restrictions in upper extremity range of motion that would prevent an individual from achieving an unhindered arm cycling motion or moving throughout a range needed to perform resistance maneuvers.
* A pressure ulcer at ischial/gluteus, trochanteric, sacral, or heel sites within the last 3 months.
* Pregnancy determined by urine testing in sexually active females.
* Imprisonment in state or federal jail or prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Postprandial insulin sensitivity | 2.5 hr
  Measured by insulin incremental area under the curve (iAUC).
Postprandial insulin sensitivity | 2.5 hr
  Measured by "ISIMatsuada" insulin sensitivity index. This index is calculated based on the ratio of blood glucose and insulin.

SECONDARY OUTCOMES:
Lipemia | 2.5 hr
  Measured by blood concentrations of triglycerides.
Carbohydrate use | 2.5 hr
  Whole-body rates of carbohydrate oxidation, as determined by open-circuit indirect calorimetry.
Fat use | 2.5 hr
  Whole-body rates of fat oxidation, as determined by open-circuit indirect calorimetry.
Fasted insulin sensitivity | Baseline
  Measured by "HOMA-2" model. This model is calculated based on the ratio of blood glucose and insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Lois Pope Life Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McMillan DW, Maher JL, Jacobs KA, Mendez AJ, Nash MS, Bilzon JLJ. Effects of Exercise Mode on Postprandial Metabolism in Humans with Chronic Paraplegia. Med Sci Sports Exerc. 2021 Jul 1;53(7):1495-1504. doi: 10.1249/MSS.0000000000002593. PMID 33433151
- [Derived] McMillan DW, Maher JL, Jacobs KA, Mendez AJ, Nash MS, Bilzon JLJ. Influence of upper-body continuous, resistance or high-intensity interval training (CRIT) on postprandial responses in persons with spinal cord injury: study protocol for a randomised controlled trial. Trials. 2019 Aug 13;20(1):497. doi: 10.1186/s13063-019-3583-1. PMID 31409383